CLINICAL TRIAL: NCT01792531
Title: The More & Less Study: A Randomized Controlled Trial Testing Different Treatment Approaches to Obesity in Preschoolers
Brief Title: The More & Less Study: A Trial Testing Different Treatment Approaches to Obesity in Preschoolers
Acronym: M&L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Paulina Nowicka, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML2012
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: children; obesity; treatment; family
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment focus - Parenting vs lifestyle (Experimental): To determine the effectiveness of two obesity treatment interventions: 1) parent training group (n=90) and 2) standard treatment with focus on lifestyle (n=90). The two treatment conditions will be evaluated with respect to child weight status (BMI SDS; primary outcome), psychosocial and metabolic health, lifestyle choices, and family functioning (secondary outcomes). This design will allow us to assess whether a program targeting only parents and focusing on parenting practices will result in better outcomes than treatment as usual emphasizing lifestyle changes.
  Interventions: Behavioral: Parent training group; Behavioral: Standard treatment with focus on lifestyle
- Length of treatment (Experimental): To understand the influence of treatment duration by comparing the effectiveness of two obesity treatment interventions: the parent training group administered for 12 wks only (n=45) and the parent training group with booster sessions which include additional booster sessions at 8-week intervals for the following year (n=45). Thus we will randomize families to either a group with booster sessions or without. This design will allow us to evaluate if prolonged care is necessary to maintain intervention effects, or if a 12-week program is equally effective.
  Interventions: Behavioral: Parent training group; Behavioral: Parent training group with booster sessions

INTERVENTIONS:
Behavioral: Parent training group — The More & Less group will focus on how to use positive parenting practices (e.g., reinforcement/encouragement, limit setting, monitoring, problem-solving, positive involvement, and emotion regulation) instead of ineffective practices (e.g., coercive behavior, negative reciprocity, escalation, and negative reinforcement). Using a parent-group approach to intervention administration, each of the twelve More & Less sessions (1.5h/wk) consist of introduction to effective parenting practices followed by a discussion and practice using role play and home practice assignments. The information and procedures will be tailored to focus on changes in the home environment, mostly related to child food habits and physical activity.
Behavioral: Standard treatment with focus on lifestyle — The treatment will be provided by local pediatricians in outpatient pediatric departments and will be based on lifestyle modifications, as recommended in the action plan for Stockholm County.
  Arms: Treatment focus - Parenting vs lifestyle
Behavioral: Parent training group with booster sessions — Parent training group with additional booster sessions at 8-week intervals for the following year.
  Arms: Length of treatment

SUMMARY:
Obesity has been shown to be resistant to treatment in adults, adolescents, and in school age children, but not during early childhood. Yet knowledge on the effectiveness of early childhood treatment programs for obesity is still very limited, preventing the widespread implementation of such programs. The overarching purpose of this study is to evaluate the effectiveness of early treatment of childhood obesity. The investigators plan to perform a carefully-designed randomized controlled trial that will evaluate different treatment options offered to families with children with obesity, organized within the healthcare system and followed up for at least 1 year post-baseline. Participants will be children aged 4-6 years (N=180) with obesity and their parents. This study will facilitate a close examination of key treatment components and mechanisms of change. Results from this study will lead to better healthcare options for obesity treatment during childhood and ultimately to the prevention of obesity later in life from a public health perspective.

DETAILED DESCRIPTION:
The proposed randomized controlled trial has four specific aims:

Specific Aim #1: PARENTING OR LIFESTYLE? To determine the effectiveness of two obesity treatment conditions: 1) parent training (n=90) and 2) treatment as usual focused on lifestyle changes (n=90). The two treatment conditions will be evaluated with respect to child weight status (BMI SDS; primary outcome), psychosocial and metabolic health, lifestyle choices, and family functioning (secondary outcomes).

Specific Aim #2: OPTIMAL LENGTH OF TREATMENT AND FOLLOW-UP? To understand the influence of treatment duration we will compare the effectiveness of the parent training program administered for 10 wks only and for 10 wks plus additional booster sessions at 8-week intervals for the following year. All groups will be followed up for at least one year post-baseline.

Specific Aim #3: TO START AT AGE 4,5 OR 6? To assess the influence of child age at the start of treatment on the treatment outcomes.

Specific Aim #4: MEDIATORS AND MODERATORS? To determine whether changes in targeted parenting skills (such as limit setting, monitoring and problem-solving) will mediate child obesity outcomes by examining all treatment groups. In addition, we will examine moderators of intervention effects (e.g. socioeconomic status (SES), parental weight status, and depression).

ELIGIBILITY:
Inclusion Criteria:

* age 4-6 years old
* obesity as defined by international cut-offs (Cole T. J. et al. BMJ, 2000).

Exclusion Criteria:

* weight affecting diseases

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) SDS | 1 year
  Measurements of children's weight and height

SECONDARY OUTCOMES:
Change in parenting practices, general and specific | 1 year
  Measured with validated questionnaires such as Child Feeding Questionnaire, Child Eating Behaviour Questionnaire and Lifestyle Behaviour Checklist. Parent's general parenting will be assessed with a questionnaire specifically developed for this study.
Change in child's dietary intake and behaviour | 1 year
  Measured using validated questionnaires such as Child Eating Behaviour Questionnaire and Food Frequency Questionnaire.
Change in child's physical activity | 1 year
  With questions about child's physical activity and screen time using Lifestyle Behaviour Checklist.
Change in family functioning | 1 year
  Using a validated questionnaire Family Assessment Device (FAD).
Change in child's metabolic health | 1 year
  Assessed by measurements of children's blood pressure, lipids, fasting glucose, insulin, and homeostasis model of insulin resistance. All these measurements are routinely assessed in all children with obesity in Stockholm. Blood tests are not required to participate in the study.
Change in parent's functioning | 1 year
  Measured by a validated questionnaire, the Beck Depression Inventory.
Waist circumference | Baseline, 3 months, 1 year
  Measured in children and parents
Change in child's functioning | 1 year
  Measured with a validated questionnaire, the Child Behaviour Checklist.
Change in socioeconomic status | 1 year
  With a questionnaire developed for this study based on routine assessments at the Child Health Care and a questionnaire used at the Oregon Social Learning Center (OSLC) for similar population (families with young children).

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Nowicka, Ph.D., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ek A, Brissman M, Nordin K, Eli K, Nowicka P. A long-term follow-up of treatment for young children with obesity: a randomized controlled trial. Int J Obes (Lond). 2023 Nov;47(11):1152-1160. doi: 10.1038/s41366-023-01373-7. Epub 2023 Oct 25. PMID 37723272
- [Derived] Sandvik P, Ek A, Eli K, Somaraki M, Bottai M, Nowicka P. Picky eating in an obesity intervention for preschool-aged children - what role does it play, and does the measurement instrument matter? Int J Behav Nutr Phys Act. 2019 Sep 3;16(1):76. doi: 10.1186/s12966-019-0845-y. PMID 31481062
- [Derived] Ek A, Lewis Chamberlain K, Sorjonen K, Hammar U, Etminan Malek M, Sandvik P, Somaraki M, Nyman J, Lindberg L, Nordin K, Ejderhamn J, Fisher PA, Chamberlain P, Marcus C, Nowicka P. A Parent Treatment Program for Preschoolers With Obesity: A Randomized Controlled Trial. Pediatrics. 2019 Aug;144(2):e20183457. doi: 10.1542/peds.2018-3457. Epub 2019 Jul 12. PMID 31300528
- [Derived] Ek A, Chamberlain KL, Ejderhamn J, Fisher PA, Marcus C, Chamberlain P, Nowicka P. The More and Less Study: a randomized controlled trial testing different approaches to treat obesity in preschoolers. BMC Public Health. 2015 Aug 1;15:735. doi: 10.1186/s12889-015-1912-1. PMID 26231850